CLINICAL TRIAL: NCT03708172
Title: rTMS and Cognitive Training for Treating Youth Depression
Brief Title: rTMS and Cognitive Training in Youth Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Z. J. Daskalakis, Chair, Temerty Centre for Therapeutic Brain Intervention, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100-2016
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Depression
Keywords: rTMS; Depression; Youth; TBS; Brain Stimulation; Electrophysiology; Imaging
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Open Label for rTMS, Double-Blinded for Cognitive Training
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS + Cognitive Training (Active Comparator): Participants will receive repetitive transcranial magnetic stimulation (rTMS) in an open label fashion. In addition, participants will receive active cognitive training (CT) which consists of completing computer-based tasks designed to enhance executive function.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation; Other: Cognitive Training
- rTMS + Sham Cognitive Training (Sham Comparator): Participants will receive repetitive transcranial magnetic stimulation (rTMS) in an open label fashion. In addition, participants will receive sham cognitive training (CT) which consists of completing computer-based tasks.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation; Other: sham Cognitive Training

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Intermittent TBS (iTBS) rTMS applied to the left Dorsolateral Prefrontal Cortex (DLPFC) + continuous TBS (cTBS) rTMS applied to the right DLPFC. The order will be counterbalanced. Administration of this treatment takes roughly 10 minutes. This treatment will be applied daily, 5 days/week, for 4 weeks.
  Other Names: MagPro rTMS Device (Magventure A/S, Farum, Denmark)
Other: Cognitive Training — Computer-based cognitive training designed to enhance executive function
  Arms: rTMS + Cognitive Training
Other: sham Cognitive Training — Computer-based inactive sham training
  Arms: rTMS + Sham Cognitive Training

SUMMARY:
Youth depression is a highly prevalent disorder with tremendous personal and societal costs. Guideline supported treatments are limited in efficacy and associated with side effects. Novel, safe, and effective treatments are sorely needed. This study will examine the biological targets, and efficacy, of cognitive training in combination with repetitive transcranial magnetic stimulation (rTMS) in non-medicated, depressed youth. If positive, the investigators will have identified an effective, safe, and acceptable alternative treatment for a population with few treatment options. Identifying biological mechanisms of response will ultimately enable clinicians to tailor individual interventions for depressed youth.

DETAILED DESCRIPTION:
Youth depression affects roughly 10% of the North American population, effecting high costs to both individuals and society at large. Unfortunately, few effective treatments exist. Antidepressant medications such as selective serotonergic reuptake inhibitors (SSRIs) are associated with side effects, and possess marginal efficacy in this age group. Black box warnings persist for antidepressants used in those under 24, owing to concerns that these medications enhance suicidal ideation in this population. While guidelines and randomized controlled trials support the use of cognitive behavior therapy (CBT) as a standalone or combination treatment for depressed youth, a large proportion of youth do not respond to either medication or psychotherapy.

The study investigators propose to examine the efficacy of repetitive transcranial magnetic stimulation (rTMS) in conjunction with cognitive training (CT) for depressed youth. rTMS delivered to the dorsolateral prefrontal cortex (DLPFC) is a safe and FDA approved treatment for adults with treatment-resistant depression, and preliminary studies suggest its safety, acceptability, and efficacy in depressed youth. Theta-burst stimulation (TBS) is a new form of rTMS that can achieve antidepressant effects in a quarter of the time of conventional rTMS. TBS is also thought to enhance neural plasticity. In this study, all participants will receive daily (5x a week on weekdays) open-label TBS. In addition, half of the participants will receive computer-based CT designed to enhance executive function, while the other half will receive placebo CT. This approach may capitalize on rTMS-induced neural plasticity, while improving depression associated executive dysfunction.

Aim:

1. to investigate the efficacy of combination cognitive training and rTMS applied to the DLPFC in youth depression, and
2. to identify biological targets and predictors of response to combined CT and rTMS intervention in youth depression

ELIGIBILITY:
Inclusion Criteria:

1. outpatients
2. between the ages of 16 and 24
3. competent to consent to study participation
4. Mini-International Neuropsychiatric Interview (MINI) confirmed diagnosis of MDD single or recurrent
5. not taking any oral medication for depression or another psychiatric indication 1-week prior to screening visit
6. HRSD-17 score of 20 and higher, to be reviewed on a case by case basis by the study psychiatrists
7. at least one failed/refused/intolerant to antidepressant trial in the current episode as determined by ATHF
8. No safety concerns endorsed on TMS Screening and Information Form

Exclusion Criteria:

1. lifetime MINI diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, delusional disorder, current psychotic symptoms, obsessive compulsive disorder, autism spectrum disorder, a history of epilepsy or any other major neurological disorder
2. diagnosis of borderline personality disorder, assessed on a case by case basis
3. at least 6 answers coded "yes" in both substance abuse and dependence sections combined, within the last 3 months as determined by MINI
4. concomitant major unstable medical illness
5. acutely suicidal or high risk for suicide as assessed by a study psychiatrist
6. not eligible to receive TMS or MRI as indicated by TMS Screening and Information Form
7. medications are considered a confound including selective serotonin reuptake inhibitors, benzodiazepines, antipsychotics, mood stabilizers, stimulants and anticonvulsants, all to be reviewed on a case by case basis
8. have failed brain stimulation in the past
9. cannot be an expert musician

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Improvement in symptom severity of depression as measured by the Hamilton Rating Scale for Depression - 17 | 5 weeks
  Hamilton Rating Scale for Depression (17-item version)
  * This scale is used to quantify the severity of symptoms of depression
  * Scale range: 0-52 (total score)
  * Lower scores indicate lower severity of depressive symptoms (i.e., better outcome)
  * Higher scores indicate higher severity of depressive symptoms (i.e., worse outcome)

SECONDARY OUTCOMES:
Improvement in self-reported symptom severity of depression as measured by the Beck Depression Inventory-II (BDI-II) | 5 weeks
  The Beck Depression Inventory-II (BDI-II) is 21-item self-report instrument intended to assess the existence and severity of symptoms of depression
  * Items are rated on a 4-point scale ranging from 0 to 3
  * Scale range: 0-63 (total score)
  * Lower scores indicate lower severity of depressive symptoms (i.e., better outcome)
  * Higher scores indicate higher severity of depressive symptoms (i.e., worse outcome)
Improvement in symptom severity of depression as measured by the Children's Depression Rating Scale, revised-version (CDRS-R) in youth under 18 years of age | 5 weeks
  The CDRS-R is a clinician-administered 17-item interview, with item ratings between 1 (=no difficulties) and 5 or 1 and 7(=clinically significant difficulties) (adding up to a total score between 17 to 113). It has been proposed, that a score of ≥40 indicates depressive symptomatology, whereas a score ≤28 was often used as indicative of remission within trials.

CONTACTS AND LOCATIONS:
Overall Officials: Z. Jeffrey Daskalakis, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Dhami P, Moreno S, Croarkin PE, Blumberger DM, Daskalakis ZJ, Farzan F. Baseline markers of cortical excitation and inhibition predict response to theta burst stimulation treatment for youth depression. Sci Rep. 2023 Nov 4;13(1):19115. doi: 10.1038/s41598-023-45107-1. PMID 37925557
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital — http://www.camh.net/research